CLINICAL TRIAL: NCT00918021
Title: Olanzapine Augmentation in Clozapine-resistant Schizophrenia: a Randomized Double-blind Study
Brief Title: Polypharmacy in Clozapine-resistant Schizophrenia
Acronym: CLOZANS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Niuvanniemi Hospital (Other)
Responsible Party: Jari Tiihonen, Professor and Chairman, Niuvanniemi Hospital, Jari Tiihonen, Professor and Chairman, Niuvanniemi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-011307-22; 0911885
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- olanzapine (B) (Active Comparator): Group B: In addition to clozapine, the participants receive their normal dosage of olanzapine (=the same as on the hospital ward) for 12 weeks, next the decreasing dosage of olanzapine for four weeks and subsequently placebo for 8 weeks.
  Interventions: Drug: olanzapine
- placebo (A) (Placebo Comparator): Group A: : In addition to clozapine the participants receive the decreasing dosage of olanzapine for four weeks, next placebo for 8 weeks, after that the increasing dosage of olanzapine for four weeks and subsequently the normal dosage of olanzapine for 8 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: olanzapine — normal dosage of olanzapine (the same dosage as on hospital ward)
  Other Names: Solazin
  Arms: olanzapine (B)
Drug: placebo — placebo
  Arms: placebo (A)

SUMMARY:
The aim of this randomized, double-blind study is to verify the hypothesis that clozapine monotherapy is as efficient as a combination of clozapine and olanzapine therapy in treatment-resistant schizophrenia.

A third of schizophrenia patients are non -responders to medications used nowadays. These patients are usually treated with clozapine, but a large proportion of patients don't recover sufficiently. Therefore, these patients are treated with combination of two or more drugs to achieve better treatment results. Until now the scientific evidence has been insufficient to assess the utility of polypharmacy.

The aim is to study during 2009 with voluntary patients, if there is any benefit of olanzapine augmentation compared with pure clozapine monotherapy. During the study the patients are not exposed to any additional intervention. The intervention in this study is just to reduce the previously used polypharmacy.

Methods: This study lasts for 24 weeks. Participants (30) are randomized in one of two alternative interventions (A or B) before the study. After 12 weeks the intervention arms cross over (from A to B and from B to A).

Group B: In addition to clozapine, the participants receive their normal dosage of olanzapine (=the same as on the hospital ward) for 12 weeks, next the decreasing dosage of olanzapine for four weeks and subsequently placebo for 8 weeks

Group A: : In addition to clozapine the participants receive the decreasing dosage of olanzapine for four weeks, next placebo for 8 weeks, after that the increasing dosage of olanzapine for four weeks and subsequently the normal dosage of olanzapine for 8 weeks

The response for the medical treatment is assessed by Clinical Global Improvement Scale (CGIS) and Global Assessment of Functioning (GAF) -scale.

The primary outcomes are GAF and modified CGIS during the parallel phase of the study (the first 12 weeks). The second phase (the last 12 weeks) of the cross-over study is used in the secondary analysis. The use of additional medication (such as benzodiazepines) is used as a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years, (adult), legally competent
* the patient is able to understand the purpose of the study and is eligible to sign the written informed consent form.
* insufficient response to the valid clozapine-olanzapine -polypharmacy
* psychotropic medication has been constant (unchangeable) during the past 2 months

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The primary outcomes are GAF and modified CGIS during the parallel phase of the study (the first 12 weeks). | 0, 12, 24 weeks

SECONDARY OUTCOMES:
The second phase (the last 12 weeks) of the cross-over study is used in the secondary analysis. The use of additional medication (such as benzodiazepines) is used as a secondary outcome measure. | 0, 12, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jari Tiihonen, MD, PhD, Principal Investigator — Niuvanniemi Hospital
Locations (1):
- Niuvanniemi Hospital, Kuopio, Finland